CLINICAL TRIAL: NCT05117554
Title: A First-in-human, Participant and Investigator-blinded, Randomized, Placebo-controlled, Single-and Multiple-Ascending Dose Study With Drug-Drug Interaction, to Investigate the Safety, Tolerability, and Pharmacokinetic Profile of AB521, in Healthy Volunteers
Brief Title: Study to Investigate the Safety, Tolerability, and Pharmacokinetic Profile With Oral AB521 in Healthy Volunteers
Acronym: ARC-14
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arcus Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ARC-14; 2021-003856-17 (EudraCT Number)
Record Dates: First submitted 2021-11-02; First posted 2021-11-11 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-05

CONDITIONS: Healthy Participants
Keywords: AB521; HIF-2α; hypoxia-inducible factor 2 alpha; Single ascending dose (SAD); Multiple ascending dose (MAD); Drug-drug interaction (DDI); casdatifan
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- SAD-casdatifan Dose 1 (Experimental): Participants will receive "Dose 1" of casdatifan orally with water under fasting conditions.
  Interventions: Drug: casdatifan
- SAD-casdatifan Dose 2 (Experimental): Participants will receive "Dose 2" of casdatifan orally with water under fasting conditions.
  Interventions: Drug: casdatifan
- SAD-casdatifan Dose 3 (Experimental): Participants will receive "Dose 3" of casdatifan orally with water under fasting conditions.
  Interventions: Drug: casdatifan
- SAD-casdatifan Dose 4 (Experimental): Participants will receive "Dose 4" of casdatifan orally with water under fasting conditions.
  Interventions: Drug: casdatifan
- SAD-Placebo (Placebo Comparator): Participants will receive matching placebo orally with water under fasting conditions.
  Interventions: Drug: Placebo
- MAD-casdatifan Dose 1 (Experimental): Participants will receive "Dose 1" of casdatifan orally with water under fasting conditions.
  Interventions: Drug: casdatifan
- MAD-casdatifan Dose 2 (Experimental): Participants will receive "Dose 2" of casdatifan orally with water under fasting conditions.
  Interventions: Drug: casdatifan
- MAD-Placebo (Placebo Comparator): Participants will receive matching placebo orally with water under fasting conditions.
  Interventions: Drug: Placebo
- DDI-casdatifan Dose + Midazolam (Experimental): Participants will receive highest safe dose level of casdatifan from MAD and midazolam orally with water under fasting conditions
  Interventions: Drug: casdatifan; Drug: Midazolam

INTERVENTIONS:
Drug: casdatifan — Capsule
  Other Names: AB521
  Arms: DDI-casdatifan Dose + Midazolam; MAD-casdatifan Dose 1; MAD-casdatifan Dose 2; SAD-casdatifan Dose 1; SAD-casdatifan Dose 2; SAD-casdatifan Dose 3; SAD-casdatifan Dose 4
Drug: Placebo — Capsule
  Arms: MAD-Placebo; SAD-Placebo
Drug: Midazolam — Syrup solution
  Arms: DDI-casdatifan Dose + Midazolam

SUMMARY:
This study will evaluate the safety and tolerability, pharmacokinetic, and pharmacodynamic profile, and drug-drug interaction (DDI) of casdatifan in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are healthy volunteers (in the opinion of the investigator) as determined by pre-study medical history, physical examination, vital signs, and 12-lead electrocardiogram (ECG)
* All clinical laboratory tests of blood and urine must be within the normal range or show no clinically relevant excursions from the normal range as judged by Principal Investigator at screening and admission.
* Screening and randomization hemoglobin ≥for males and females is as follows:

  * SAD: male and female hemoglobin level ≥ 12.5 grams/ deciliters (g/dL) (7.7 millimoles/liters [mmol/L])
  * MAD and DDI: male hemoglobin level ≥ 14.2 g/dL (8.8 mmol/L) and female hemoglobin level ≥ 12.5 g/dL (7.7 mmol/L).
* Participants should have adequate peripheral venous access.
* Body weight of 45 kilograms (kg) or greater and body mass index within the range of 18 to 32 kg/meters squared (m^2) (inclusive)
* Male participants must be vasectomized and have been vasectomized for at least 3 months prior to screening visit with confirmed history of azoospermia subsequent to the vasectomy procedure
* Contraceptive use should be consistent with local regulations

Exclusion Criteria:

* Has any (acute or chronic [including severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection]) medical or psychiatric condition that, in the opinion of the investigator, could jeopardize or would compromise the study participant's ability to participate in this study
* Has history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, hematological, cerebrovascular, neurological, or other major disorders capable of significantly altering the absorption, metabolism, or elimination of investigational drug; constituting a risk when taking the study intervention; or interfering with the interpretation of data in the opinion of the investigator
* Abnormal blood pressure (BP) or pulse measurements at the Screening Visit or Day -2/-1 (Admission) in a supine position after 5 minutes of rest as follows: mean systolic BP ≥139 millimeters of mercury (mm Hg) or mean diastolic BP ≥89 mm Hg; mean pulse < 40 beats per minute (bpm) or > 100 bpm.
* Liver enzyme test results: Alanine aminotransferase, aspartate aminotransferase, bilirubin, or alkaline phosphatase >1.0x the upper limit of normal
* Current or chronic history of liver disease or known hepatic or biliary abnormalities
* Has 12-lead electrocardiogram with changes considered to be clinically significant at the Screening Visit or day of admission

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2021-11-09 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-02-17 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) | Up to 21.5 Weeks
Number of Participants With Abnormal Changes From Baseline in Laboratory Parameter Values | Baseline; Up to 21.5 Weeks
Number of Participants With Abnormal Changes from Baseline in Vital Sign Values | Baseline; Up to 21.5 Weeks
Maximum Observed Plasma Concentration (Cmax) of casdatifan | multiple timepoints up to approximately 21.5 Weeks
Area Under the Plasma Concentration Time Curve From Hour 0 to the Last Sample With Measurable Plasma Concentrations (AUClast) of casdatifan | multiple timepoints up to approximately 21.5 Weeks
Time of Occurrence of Cmax (tmax) of casdatifan | multiple timepoints up to approximately 21.5 Weeks
Apparent Terminal Elimination Rate Constant (λz) of casdatifan | multiple timepoints up to approximately 21.5 Weeks
Terminal Half-Life (t1/2) of casdatifan | multiple timepoints up to approximately 21.5 Weeks
Area Under the Plasma Concentration Time Curve From Hour 0 to Infinity (AUCinf) of casdatifan | multiple timepoints up to approximately 21.5 Weeks
Apparent Volume of Distribution of casdatifan | multiple timepoints up to approximately 21.5 Weeks
Apparent Total Body Clearance of casdatifan | multiple timepoints up to approximately 21.5 Weeks

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of midazolam and 1 hydroxymidazolam | multiple timepoints up to approximately 21.5 Weeks
Area Under the Plasma Concentration Time Curve From Hour 0 to the Last Sample With Measurable Plasma Concentrations (AUClast) of midazolam and 1 hydroxymidazolam | multiple timepoints up to approximately 21.5 Weeks
Time of Occurrence of Cmax (tmax) of midazolam and 1 hydroxymidazolam | multiple timepoints up to approximately 21.5 Weeks
Apparent Terminal Elimination Rate Constant (λz) of midazolam and 1 hydroxymidazolam | multiple timepoints up to approximately 21.5 Weeks
Terminal Half-Life (t1/2) of midazolam and 1 hydroxymidazolam | multiple timepoints up to approximately 21.5 Weeks
Area Under the Plasma Concentration Time Curve From Hour 0 to Infinity (AUCinf) of midazolam and 1 hydroxymidazolam | multiple timepoints up to approximately 21.5 Weeks
Apparent Volume of Distribution of midazolam and 1 hydroxymidazolam | multiple timepoints up to approximately 21.5 Weeks
Apparent Total Body Clearance of midazolam and 1 hydroxymidazolam | multiple timepoints up to approximately 21.5 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Arcus Biosciences, Inc.
Locations (1):
- Investigational Site, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Arcus will provide access to individual de-identified participant data and related study documents (e.g., protocol, Statistical Analysis Plan [SAP], Clinical Study Report [CSR]) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions.
  For more information, please visit our website.
Supporting Information: Study Protocol, SAP, CSR
URL: https://trials.arcusbio.com/our-transparency-policy

REFERENCES:
- See also: ARC-14 - Public website — https://trials.arcusbio.com/study/?id=ARC-14